CLINICAL TRIAL: NCT03583047
Title: Intracoronary Profile of Inflammation, Oxidative Stress and Endothelial Progenitor Cells (EPCs) in the Prognosis of Endothelial Dysfunction, Stent Re-stenosis and Cardiovascular Events in Population With Acute Coronary Syndrome.
Brief Title: Intracoronary Features in the Prognosis of Endothelial Dysfunction and MACES in Population With Acute Coronary Syndrome
Acronym: iphoneSPACE
Status: Completed | Type: Observational
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Juan Antonio Suárez Cuenca, Principal Investigator, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Other Study IDs: CONS0008-2014-1
Record Dates: First submitted 2018-06-04; First posted 2018-07-11 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Endothelial Dysfunction; Cardiovascular Risk Factor; Coronary Syndrome, Acute
Keywords: MACE; EPCs; Cardiovascular risk; Endothelial dysfunction; Prognosis
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — total blood blood serum, and blood plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary Artery Disease (CAD) is common in Mexico, while morbidity and mortality is high. Drug therapy can relieve angina pain and stabilize plaque, but it is not able to re-flow a coronary artery. Balloon angioplasty and/or stent placement, re-establishes coronary blood flow; however, the risk of re-stenosis and/or development of new coronary events remains latent. Endothelial damage, reflected by the degree of endothelial dysfunction, inflammation and oxidative stress, promotes atherogenesis, which plays a central role in the pathophysiology of CAD. These mechanisms have been studied in animal models; however, it is widely unknown whether it influences the coronary circulation in humans. Therefore the present study explores the impact of an intracoronary profile of biomarkers of endothelial dysfunction, inflammation and oxidative stress on the prognosis of coronary remodeling and new adverse cardiovascular events in patients with chronic stable coronary syndrome undergoing angioplasty and stent placement.

DETAILED DESCRIPTION:
Study design: Observational, longitudinal, analytic and prospective cohort study.

.With the Ethics and institutional investigation Committee acceptance, patients with stable coronary plaque or post-infarct angina with indicated coronary angiography and stent placement, from the Hemodynamic Unit from the National Medical Center "20 de Noviembre" of the Institute of Security and Social Services of State Workers (ISSSTE) are invited to participate. Patients who agree to participate in the study sign the informed consent. The independent variables will be the coronary profile components (oxidative stress, inflammation and endothelial disfunction biomarkers) and the consequence variables (dependent) will be the coronary and/or stent remodeling during the post-angioplasty with stent placement monitoring, Major Adverse Cardiovascular Events (MACE) during the post-angioplasty with stent placement monitoring period.

Clinical data:

to homogenize the study population respect to potentially confusing variables, information about sex, age, body mass index, vital signs. lipid profile. co-morbility presence like systemic arterial hypertension, diabetes mellitus, metabolic syndrome, drugs and troponin determination for stratify the acute coronaropathy.

Coronary Catheterization and sampling. The coronary catheterization (angioplasty with stent placement) is made under medical indication.

-Coronary catheterism: Is made in the hemodynamic laboratory. Asepsis, antisepsis and local anesthesia are performed in the intravascular approach area.

ELIGIBILITY:
Inclusion Criteria:

* Coronary syndrome patients
* Patients with Endothelial dysfunction

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Ischemic patients who are submitted to a percutaneous coronary intervention.
  * Atherosclerotic patients with coronary stent.
  * All the patients included are from the hospital "20 de noviembre, ISSSTE" in Mexico City.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Development of any Major Adverse Cardiovascular Event (MACE) | 3 months
  Development of any MACE (a combination of major cardiovascular events, including death, heart failure, post-infarction angina, or new myocardial infarction) during a 3 months follow-up after angioplasty and stent placement.

SECONDARY OUTCOMES:
Development of any Major Adverse Cardiovascular Event (MACE) | 6 months
  Development of any MACE (A combination of any major cardiovascular events, including death, heart failure, post-infarction angina or new myocardial infarction) during a 6 months follow up after angioplasty and stent placement

CONTACTS AND LOCATIONS:
Overall Officials: Juan A. Suárez-Cuenca, Ph.D, Principal Investigator — Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Locations (1):
- National Medical Center "20 de Noviembre", ISSSTE, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No